CLINICAL TRIAL: NCT06497244
Title: Evaluation of the Effect of Micro-osteoperforation on the Rate of Bone Anchored Molar Distalization: a Split-mouth Randomized Controlled Clinical Trial
Brief Title: Evaluation of the Effect of Micro-osteoperforation on the Rate of Bone Anchored Molar Distalization
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohamed essam, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MOPD-CU-2022-11-15
Record Dates: First submitted 2024-06-24; First posted 2024-07-11 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Microosteoperforations

STUDY DESIGN:
Intervention Model Description: Subjects will receive MOPs randomly to either the left or right maxillary molar buccal alveolar regions. MOPs will be performed at the first day of the distalization treatment (T0) and will repeated every 2 months.
Who Masked: Outcomes Assessor
Masking Description: The first assessor will perform the digital models & CBCT measurements blindly for each patient. The second assessor will perform the same measurements blindly to calculate the inter-observer error
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- micro osteo-perforation side (Experimental): the patient will receive micro osteo-perforation in one side Computer generated random numbers will generated using Microsoft Office Excel sheet by a person who was not involved in the clinical trial. Because of the split mouth design, the right sides of patients will randomly be assigned to one of the two groups (MOPs or control). Then, the left sides will automatically be assigned to the alternative group.
  Interventions: Procedure: micro osteo-perforation
- no micro osteo-perforation side (No Intervention): the other side without micro osteo-perforation

INTERVENTIONS:
Procedure: micro osteo-perforation — the patient will receive miniscrew micro osteo-perforation in one side every month with molar distalization and the other side the distalization without micro osteo-perforation
  Arms: micro osteo-perforation side

SUMMARY:
The primary aim of the current study was to evaluate three dimensionally, using digital models and cone beam computed tomography imaging, the effect of micro-osteoperforations on the rate of tooth movement in the first molar distalization.

DETAILED DESCRIPTION:
The design of this randomized controlled clinical trial is a parallel group, two arms trial

* Preparatory phase

  * Self-drilling mini-screws will be placed buccally between upper 2nd premolar and 1st molar bilaterally in the last NiTi wire insertion visit.
  * After the completion of levelling and alignment phase an intra oral scan will be made for the upper arch and a rigid stainless-steel retraction arch wire 0.017" x 0.025" will be inserted.
  * The patient will then be referred to the radiology center and a pre-retraction cone beam computed tomography (CBCT) image will be taken for the maxillary arch (T0).
* Experimental phase

  * Subjects will receive MOPs randomly to either the left or right maxillary molar buccal alveolar regions. MOPs will be performed at the first day of the distalization treatment (T0) and will repeated every 2 months.
  * Molar distalization will started immediately after performing the MOPs using sliding jig distalizer.
  * The force will be applied to the mini-screw with the sliding jig mechanics on average 300 gm using Nickel-titanium closing coil springs.
  * Before leaving the clinic, the patient will be asked to:
  * Use chlorhexidine three times per day for 3 days after MOP applications.
  * avoid using pain killers (except Panadol when needed).
  * fill in a Numeric pain rating scale.
* Follow up phase

  * Follow up visits will be scheduled every 4 weeks for reactivation coil spring and check TADs stability.
  * An intra oral scan for the upper arch will made every visit.
  * The study time will be continued for 6 months (T1, T2, T3, T4, T5, T6).
  * The same technique of MOP will be repeated after 2 and 4 months of follow up (T2,T4).
  * After 6 months of follow up, the final dental model will made, and the patient will be referred to the same radiology center to acquire the post-distalization CBCT.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients
2. Skeletal Class I or mild Class II relationship
3. Dental class II bilaterally (non-extraction cases)
4. Full permanent dentition including 2nd maxillary molars
5. Good oral hygiene
6. Medically free

Exclusion Criteria:

1. Systemic diseases that may interfere with the treatment
2. Use of any medications that might have affected the biology of tooth movement
3. unilateral Class II molar relationship
4. extreme skeletal Class II relationship (ANB >7°)
5. periodontal disease or alveolar bone loss
6. Patients with dental anomalies in maxillary 1st molar

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
rate of molar distalization | 6 months
  Incremental rate of molar distalization every month by intra oral scan superimposition
total molar distalization distance by mm between T6 and T0 | 6 months
  Total distance moved by the molar after 6 months by intra oral scan superimposition and measure the linear difference in position 1st molar between T6 and T0 by mm

SECONDARY OUTCOMES:
The effect of MOPs on Maxillary 1st molar tipping by degrees between T6 and T0 | 6 months
  comparing the pre- & post- distalization CBCT and measure the angular change in the 1st molar long axis tipping by degree between T6 and T0
The effect of MOPs on Maxillary 1st molar rotation by degrees between T6 and T0 | 6 months
  comparing the pre- & post- distalization digital models and CBCT and measure the angular change in the 1st molar long axis rotation by degree between T6 and T0
The effect of MOPs on Maxillary 1st molar vertical movement by mm between T6 and T0 | 6 months
  comparing the pre- & post- distalization CBCT and measure the linear change in the 1st molar vertical position by mm between T6 and T0
The effect of MOPs on 1st molar root resorption level by mm between T6 and T0 | 6 months
  comparing the pre- & post- distalization CBCT and measure the amount of root resorption of 1st molar roots by mm between T6 and T0
Detecting any Pain or discomfort caused by the micro-osteoperforations using Numeric pain rating scale | 1 week
  using Numeric Pain Rating Scale filled by the patient with minimum value is zero and maximum value 10 (the higher score mean worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Abdou, professor, Study Chair — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No